CLINICAL TRIAL: NCT01144546
Title: Passive Leg Raising Test to Predict Hypotension During Induction of Anesthesia in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Yunseok Jeon, MD., Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-0809-037-256
Record Dates: First submitted 2010-06-08; First posted 2010-06-15 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2010-06

CONDITIONS: Ischemic Heart Disease; Cardiac Valve Disease
Keywords: Passive leg raising; FloTrac/Vigileo; Anesthesia hypotension
MeSH Terms: conditions — Myocardial Ischemia; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Passive Leg Raising (Experimental): elevation of both legs to a 45 degrees for about 1-2 minute before anesthesia induction
  Interventions: Procedure: passive leg raising (45 degree leg elevation for 1-2 min)

INTERVENTIONS:
Procedure: passive leg raising (45 degree leg elevation for 1-2 min) — the patient's trunk was elevated 45 degrees for the first set of measurements. Then, the lower limbs were raised to a 45° angle while the patient's trunk was lowered to a supine position to measure peak CO (usually within 1-2 min)
  Other Names: PLR

SUMMARY:
Hypotension frequently occurs during anesthesia induction. Preload decrease by anesthetics was often considered as one of main causes for this hypotension. However, the studies on this topic have been lacking. Dynamic preload indices are more suitable than static preload indices to predict the effect of preload changes. And, recently, passive leg raising test showed successful results to predict fluid responsiveness in patient with spontaneous ventilation.

The investigators hypothesized that hypotension after induction of anesthesia is caused by decrease of preload by anesthetics and passive leg raising test could predict this hypotension. In this study, the investigators will try to evaluate whether passive leg raising induced hemodynamic changes could predict hypotension during anesthesia induction.

DETAILED DESCRIPTION:
In this randomized controlled clinical trial, the investigators hypothesized that passive leg raising induced changes in hemodynamic parameters could predict the hypotension during anesthesia induction. To evaluate this, before anesthesia, the investigators will conduct passive leg raising test. At first, the patient's trunk was elevated 45 degrees for the first set of measurements. Then, the lower limbs were raised to a 45° angle while the patient's trunk was lowered to a supine position to measure peak CO (usually within 1-2 min). Hemodynamic profiles planned to be measured are mean arterial pressure, heart rate, cardiac index, stoke volume and stroke volume variation. After this, the occurrence of hypotension (systolic blood pressure < 90mmHg or mean arterial pressure decrease > 30% of baseline) will be recorded during the time from anesthesia induction to surgical skin incision. Hypotension will be treated by a standardized method. If heart rate (HR) is less than 70 beats/min, 5mg of ephedrine will be administered and if HR is greater than 70 beats/min, 30 mcg of phenylephrine will be administered. This will repeated until hypotension subsided. Refractory hypotension will be defined as continuous hypotension despite the total infused dose of ephedrine > 0.5 mg/kg or phenylephrine > 4 mcg/kg. The ability to predict hypotension and refractory hypotension during anesthesia induction by passive leg raising test will be evaluated by receiver operating characteristic curve analysis.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing elective cardiac surgery

Exclusion Criteria:

* arrhythmias
* documented peripheral artery disease
* severe pulmonary disease
* heart failure
* unstable angina
* preoperative use of inotropics or mechanical assist device
* use of angiotensin converting enzyme inhibitors
* expected intubation difficulty or gastric reflux disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-08; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The area under ROC curve to predict hypotension and refractory hypotension | 30 min around passive leg raising test
  area under ROC curve of HR, SV, SVV, and CI changes during PLR to predict hypotension and refractory hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, M.D, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea